CLINICAL TRIAL: NCT03204305
Title: Brain Imaging of Cannabinoid Receptors in Women
Brief Title: Brain Imaging of Cannabinoid Receptors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00101744; R21DA043963 (NIH)
Record Dates: First submitted 2017-05-30; First posted 2017-07-02 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Cannabis Use Disorder; Cannabis Dependence, Continuous
Keywords: Marijuana; cannabis; cannabinoid receptor
MeSH Terms: conditions — Marijuana Abuse | interventions — 4-cyano-1-(2,4-dichlorophenyl)-5-(4-methoxyphenyl)-N-(piperidin-1-yl)-1H-pyrazole-3-carboxamide; nabiximols

STUDY DESIGN:
Intervention Model Description: Two groups will be recruited. Female cannabis users and nonusers.
Who Masked: Participant
Masking Description: Cannabis THC content (dose) is masked for participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabis users (Active Comparator): Smoked Cannabis plant material (0 and 25 mg THC) will be administered to volunteers who are regular cannabis users. Cannabis users will also complete a PET scan where 20 millicurie of 11C-OMAR
  Interventions: Drug: 11C-OMAR; Drug: Cannabis
- Nonuser controls (Active Comparator): No cannabis administration. Non-user controls will complete a PET scan where 20 millicuries of 11C-OMAR
  Interventions: Drug: 11C-OMAR

INTERVENTIONS:
Drug: 11C-OMAR — 11C-OMAR is a PET radiotracer that binds to cannabinoid type 1 receptors (CB1R). It is an analog of the CB1R antagonist/inverse agonist rimonabant. 11C-OMAR was developed, synthesized and validated for inhuman use at the Johns Hopkins University PET center.
  Other Names: JHU75528
Drug: Cannabis — Cannabis will be administered to cannabis users. Doses include 0 and 25 mg THC.
  Other Names: Marijuana
  Arms: Cannabis users

SUMMARY:
All participants will be healthy volunteers and all procedures will be completed for research purposes only. Two groups will be recruited, females who use cannabis (marijuana, MJ), and female who do not use cannabis (controls). Female MJ users will be enrolled in a protocol that includes an outpatient drug administration session and a 4-day/3-night inpatient stay on the Johns Hopkins Bayview Clinical Research Unit (CRU). During outpatient visits, MJ users will have an MRI, and complete MJ self-administration and cognitive performance sessions. MJ users will then reside on the CRU,and complete MJ abstinence, and self-report instruments for withdrawal discomfort. A positron emission tomography (PET) scan of brain cannabinoid type 1 receptors will also be completed. Non-users will complete MRI, PET imaging and cognitive testing under an outpatient protocol (no MJ administration).

DETAILED DESCRIPTION:
The primary goals of this project are to examine whether use of cannabis alters brain cannabinoid type 1 receptor (CB1R) availability in females, and if severity of cannabis withdrawal is correlated with CB1 receptor availability. CB1R are widely distributed in the human brain and can be quantified using PET imaging with the radiotracer 11C-OMAR (Carbon-11-OMAR). The effects MJ use on brain CB1R have not been studied in females. The current study will enroll 10 female MJ users in an inpatient protocol that includes administration of smoked MJ, followed by monitored abstinence with daily behavioral assessments, and PET imaging with 11C-OMAR. PET data will collected in 10 matched controls for comparison. The proposed study is an important first step to determine whether localized CB1R changes in female MJ users help explain, and provide a neurobiological target for intervention. Results will increase knowledge of cannabinoid mechanisms of cannabis use and severity of dependence in females, an understudied population.

ELIGIBILITY:
* Female, healthy adult volunteers who are either MJ users and nonusers (controls)
* 18-45 years of age
* serum creatinine and hepatic enzymes (AST, ALT) must be within the normal limits
* Women of child bearing potential must meet one of the following three criteria:

  1. negative pregnancy test by serum pregnancy test 2 .Following a reliable method of birth control 3. Agreeing to follow a reliable method of birth control during the study and for 1 month following all study procedures

Additional inclusion criteria for MJ users

* Regular MJ use
* present MJ positive urine
* meet Diagnostic and Statistical Manual, version 5 (DSM-5) criteria for cannabis use disorder (CUD)

Additional inclusion non-users

* report no MJ use
* present a MJ-negative urine

Exclusion Criteria:

* < 5th grade reading level
* Current Diagnostic and Statistical Manual, version 5 (DSM-5) psychiatric disorder;
* Current DSM-5 alcohol or substance use disorder (excluding MJ or nicotine)
* Recent Illicit drug use or positive drug test
* Using MJ under the guidance of MD;
* History of seizures, closed head trauma;
* unstable hypertension;
* conditions preventing magnetic resonance imaging (MRI) such as implanted metal, claustrophobia, or anatomical abnormalities (e.g., enlarged ventricles, brain lesions);
* Use of medications or herbal supplements which may be counter indicated as determined by study physician
* Have had exposure to ionizing radiation that in combination with the study's estimated radiation exposure would result in a cumulative exposure that exceeds recommended exposure limits of 5 rem per year.
* Presence or history of drug allergy, or allergic disease diagnosed and treated by a physician.
* any serious medical condition in whom participation is contraindicated.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise Weerts, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 participants (8 females, 7 males) did not start, but were historical controls included for data analysis
Groups:
- Female Cannabis Users: Females with cannabis use disorder (CUD): reported using cannabis on average ≥ 25 days per month in the past 3 months, positive test for cannabis on a urine screen, met DSM-V criteria for moderate or severe CUD, and reported ≥ 2 cannabis withdrawal symptoms during a past cannabis abstinence period.
- Female Healthy Nonuser Controls: Female healthy controls (nonusers): no cannabis use for ≥ 12 months, ≤ 5 lifetime cannabis uses, negative urine test for cannabis
- Female Non-user Healthy Historical Controls: Female non-users who were not enrolled in the study but were collapsed into the same category as contemporary controls (n = 2) bringing total number of female non-user healthy controls to 10.
- Male Healthy Historical Controls: Male healthy historical controls (nonusers) who were not enrolled in the study but were used for gender comparison
Period: Overall Study
Arm/Group | Female Cannabis Users | Female Healthy Nonuser Controls | Female Non-user Healthy Historical Controls | Male Healthy Historical Controls
Started | 21 | 7 | 8 | 7
Completed | 10 | 2 | 8 | 7
Not Completed | 11 | 5 | 0 | 0
Not completed — Lost to Follow-up | 6 | 4 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — failure to place arterial line | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 21 female cannabis users and 7 female healthy control nonusers enrolled. Of these, 10 of the female cannabis users and 2 healthy control female nonusers completed the full protocol and were included in the analysis. Due to low recruitment for healthy controls, 8 historical female healthy controls were included in analysis. We also conducted an analysis that compared all female controls (n=10; 2 healthy controls and 8 matched historical controls) with male historical controls.
Groups:
- Female Cannabis Users With CUD: Smoked Cannabis plant material (0 and 25 mg THC) will be administered to volunteers who are regular cannabis users. Cannabis users will also complete a PET scan where 20 millicurie of 11C-OMAR
  11C-OMAR: 11C-OMAR is a PET radiotracer that binds to cannabinoid type 1 receptors (CB1R). It is an analog of the CB1R antagonist/inverse agonist rimonabant. 11C-OMAR was developed, synthesized and validated for inhuman use at the Johns Hopkins University PET center.
  Cannabis: Cannabis will be administered to cannabis users. Doses include 0 and 25 mg THC.
- Nonuser Female Healthy Controls (Contemporary and Historical): No cannabis administration. Non-user controls will complete a PET scan where 20 millicuries of 11C-OMAR.
  11C-OMAR: 11C-OMAR is a PET radiotracer that binds to cannabinoid type 1 receptors (CB1R). It is an analog of the CB1R antagonist/inverse agonist rimonabant. 11C-OMAR was developed, synthesized and validated for inhuman use at the Johns Hopkins University PET center.
  Contemporary and historical female non-user healthy controls were collapsed into one group due to low enrollment of contemporary healthy controls.
- Male Non-user Historical Controls: Historical male non-user healthy controls used for comparison
- Total: Total of all reporting groups
Arm/Group | Female Cannabis Users With CUD | Nonuser Female Healthy Controls (Contemporary and Historical) | Male Non-user Historical Controls | Total
Number analyzed (Participants) | 10 | 10 | 7 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (2.7) | 25.5 (5.0) | 29.6 (6.9) | 25.7 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 0 | 20
  Male | 0 | 0 | 7 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 5 | 11
  White | 4 | 9 | 1 | 14
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Age of first cannabis use [Mean (Standard Deviation); unit: years] — Population: Only 10 participants were cannabis users (healthy controls had used cannabis ≤ 5 times in lifetime); therefore, "age of first cannabis use" data was only collected for the group of cannabis users.
  years
    number analyzed (Participants) | 10 | 0 | 0 | 10
    (all) | 15.3 (3.0) |  |  | 15.3 (3.0)
Years of cannabis use [Mean (Standard Deviation); unit: years] — Population: Only 10 participants were cannabis users (healthy controls had used cannabis ≤ 5 times in lifetime); therefore, "years of cannabis use" only applies to the group of cannabis users.
  years
    number analyzed (Participants) | 10 | 0 | 0 | 10
    (all) | 7.9 (4.3) |  |  | 7.9 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Distribution Volume (VT)
Description: Distribution Volume (VT) is the quantification of 11C-OMAR binding to the CB1R; Per our statistical plan we examined VT for eight volumes of interest in the brain (ventral striatum, amygdala, putamen, cingulate, globus pallidus, insula, frontal cortex, and hippocampus) as well as the composite VT for the brain. The unit of measure is mL/cm^3.
Time Frame: Collected during 90-min PET study
Population: Nonuser female healthy controls group includes 2 contemporary female controls and 8 historical female controls.
Measure: Mean (Standard Error); unit: mL/cm^3
Groups:
- Nonuser Female Healthy Controls: No cannabis administration. Non-user controls will complete a PET scan where 20 millicuries of 11C-OMAR
  11C-OMAR: 11C-OMAR is a PET radiotracer that binds to cannabinoid type 1 receptors (CB1R). It is an analog of the CB1R antagonist/inverse agonist rimonabant. 11C-OMAR was developed, synthesized and validated for inhuman use at the Johns Hopkins University PET center.
- Historical Non-user Male Healthy Controls: Healthy, non-user historical male controls
Arm/Group | Cannabis Users | Nonuser Female Healthy Controls | Historical Non-user Male Healthy Controls
Number analyzed (Participants) | 10 | 10 | 7
mL/cm^3
  Amygdala VT | 1.27 (0.19) | 1.54 (0.29) | 1.14 (0.18)
  Cingulate VT | 1.31 (0.2) | 1.56 (0.27) | 1.19 (0.16)
  Frontal lobe VT | 1.29 (0.19) | 1.51 (0.26) | 1.18 (0.16)
  Globus Pall VT | 1.77 (0.29) | 1.87 (0.35) | 1.38 (0.24)
  Hippocampus VT | 1.28 (0.20) | 1.54 (0.29) | 1.19 (0.19)
  Insula VT | 1.37 (0.21) | 1.62 (0.28) | 1.24 (0.18)
  Putamen VT | 1.52 (0.21) | 1.69 (0.29) | 1.31 (0.19)
  Ventral straitum VT | 1.36 (0.22) | 1.52 (0.26) | 1.21 (0.18)
  Composite VT | 1.27 (0.19) | 1.45 (0.24) | 1.15 (0.16)
Statistical Analysis 1: Comparison: Cannabis Users vs Nonuser Female Healthy Controls; VT in the 8 volumes of interest were analyzed using linear regression model group coded encoded as a dummy variable [1=females cannabis users; 2= female healthy controls], age as a covariate, and VT for VOIs (ventral striatum, amygdala, putamen, cingulate, globus pallidus, insula, frontal cortex, and hippocampus) as dependent variables, followed by post hoc Tukey's HSD between between groups; Test type: Superiority; p = 0.02, t-test, 2 sided — p < 0.05 for all analyses. Bonferroni corrections were made to reduce family-wise error rate; Composite VT was compared using independent t-tests; t-test = -2.51
Statistical Analysis 2: Comparison: Cannabis Users vs Nonuser Female Healthy Controls; Test type: Superiority; p = 0.03, t-test, 2 sided; t-test = -2.36
Statistical Analysis 3: Comparison: Cannabis Users vs Nonuser Female Healthy Controls; Test type: Superiority; p = 0.03, t-test, 2 sided; t-test = -2.35
Statistical Analysis 4: Comparison: Cannabis Users vs Nonuser Female Healthy Controls; Test type: Superiority; p = 0.04, t-test, 2 sided; t-test = -2.23

2. Secondary Outcome: Peak Change From Baseline Marijuana Withdrawal Discomfort Score
Description: Marijuana withdrawal discomfort will be self-reported using the marijuana withdrawal checklist, available via PhenXToolkit.org. Items are: depressed mood, irritability, nervousness/anxiety, restlessness, increased aggression, increased anger, violent outbursts, nausea, decreased appetite, stomach pain, shakiness, sweating, sleep difficulty, strange/wild dreams, craving to smoke cannabis, diarrhea/loose stools, dizziness, muscle spasms/aches, hiccups, stuffy nose, feverish feeling, hot flashes, chills, increased appetite, headaches, fatigue/tiredness, yawning, difficulty concentrating, general physical discomfort, and other. Each item is rated as 0=none, 1=mild, 2=moderate, or 3=severe. A sum score is calculated from items that are valid, reliable cannabis withdrawal symptoms (Budney et al, 2003, Journal of Abnormal Psychology,112(3): 393-402). A higher score represents more severe withdrawal. Scores range from 0-36.
Time Frame: Up to 5 days
Population: Females with CUD who completed cannabis administration sessions 1 and 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cannabis Users: Smoked Cannabis plant material (0 and 25 mg THC) will be administered to volunteers who are regular cannabis users. They then will undergo an inpatient period of abstinence for 3 days.
  Cannabis: Cannabis will be administered to cannabis users. Doses include 0 and 25 mg THC.
Arm/Group | Cannabis Users
Number analyzed (Participants) | 14
score on a scale
  Marijuana Withdrawal Discomfort Score: Score Pre Cannabis Administration session 2 | 2.30 (2.26)
  Marijuana Withdrawal Discomfort Score: Peak score during 3 day Inpatient abstinence period | 4.80 (3.85)
Statistical Analysis 1: Comparison: Cannabis Users; Test type: Superiority; p = 0.03, t-test, 2 sided; t test = -2.52

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse event data not available for historical control males or historical control females.
Groups:
- Females With Cannabis Use Disorder: Smoked Cannabis plant material (0 and 25 mg THC) will be administered to volunteers who are regular cannabis users. Cannabis users will also complete a PET scan.
- Nonuser Female Healthy Controls: No cannabis administration. Non-user controls will complete a PET scan.
- Historical Female Controls: Historical female controls who completed a PET scan
- Historical Male Controls: Historical male controls who completed a PET scan
Arm/Group | Females With Cannabis Use Disorder | Nonuser Female Healthy Controls | Historical Female Controls | Historical Male Controls
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/7 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/7 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/21 | 0/7 | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT03204305/Prot_SAP_000.pdf